CLINICAL TRIAL: NCT02656719
Title: Comparison Between Bronchoscopy and Real- Time Ultrasound Guided Percutaneous Dilatational Tracheostomy for Safety, Complications and Efficiency in Critically Ill Patient
Brief Title: Comparison Between Bronchoscopy and Real- Time Ultrasound Guided Percutaneous Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aykut Saritas (Other)
Collaborators: Prof.Dr.A.İlhan Özdemir State Hospital (Other)
Responsible Party: Sponsor-Investigator, Aykut Saritas, principal investigator, Tepecik Training and Research Hospital
Organization: Tepecik Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1
Record Dates: First submitted 2016-01-05; First posted 2016-01-15 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Tracheostomy Complications
Keywords: tracheostomy; complications; ultrasound; bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Ultrasound guided percutaneous tracheostomy
  Interventions: Device: Ultrasound guided percutaneous tracheostomy
- Bronchoscopy (Active Comparator): Bronchoscopy guided percutaneous tracheostomy
  Interventions: Device: Bronchoscopy guided percutaneous tracheostomy

INTERVENTIONS:
Device: Ultrasound guided percutaneous tracheostomy — Ultrasound guided percutaneous tracheostomy
  Arms: Ultrasound
Device: Bronchoscopy guided percutaneous tracheostomy — Bronchoscopy guided percutaneous tracheostomy
  Arms: Bronchoscopy

SUMMARY:
Trial is a randomized study to compare between ultrasound guided percutaneous tracheostomy and bronchoscopy guided percutaneous tracheostomy.

DETAILED DESCRIPTION:
Trial is a randomized study to compare between ultrasound guided percutaneous tracheostomy and bronchoscopy guided percutaneous tracheostomy.

Patients will be randomly assigned to be submitted to evaluate safety, complication rates, easy to perform , clinical outcomes and effectivity.

ELIGIBILITY:
Inclusion Criteria:

* All intubated and mechanically ventilated patients indicated for a tracheostomy

Exclusion Criteria:

* Patients with tracheal or neck abnormalities, soft tissue infection in the neck, neck surgery history, oxygenation problems , coagulation disorders or coagulation parameter changes and those requiring urgent or surgery patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
procedure failure of ultrasound to provide this anatomical information and ease of perform | During percutaneous tracheostomy an expected average time 20 minutes
  occurence of a major complications: bleeding, subcutaneous emphysema, oesophageal perforation, number of applied needle interventions, procedure duration, cardiorespiratory arrest

SECONDARY OUTCOMES:
procedure time | during percutaneous tracheostomy ( average expected time 20 minutes)
  the procedure duration was taken as the time that elapsed from the placement of the needle to the placement of the tracheostomy cannula.
Pneumothorax | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Pneumothorax due to the percutaneous tracheostomy detected by clinical examination during the procedure or chest x-ray after the procedure.
Tracheal posterior wall injury | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Tracheal posterior wall injury as detected by bronchoscopy after the procedure
Accidental decannulation | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Accidental decannulation after the procedure during Hospital stay
Cardiorespiratory arrest | during percutaneous tracheostomy an expected average of 20 minutes
  Cardiorespiratory arrest due to percutaneous tracheostomy
Minor bleeding | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Haemorrhage that could not be stopped by sponge wrapping the stoma after the procedure and/or blood coming with aspiration inside the tracheostomy tube was defined as minor bleeding
Major bleeding | During the procedure an expected average of 20 minutes
  Continuous haemorrhage from the stoma and/or from the trachea with aspiration despite compresses was defined as a major haemorrhage.

OTHER OUTCOMES:
Hypoxemia | During percutaneous tracheostomy an expected average of 20 minutes
  Drop in peripheral oxygen saturation < 90% for more than 2 minutes as measured by pulse oximeter during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Aykut Saritas, MD, Principal Investigator — İzmir Tepecik Training and Research Hospital; muhammed murat kurnaz, MD, Study Chair — Prof.Dr.A.İlhan Ozdemir State hospital Giresun

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ravi PR, Vijay MN. Real time ultrasound-guided percutaneous tracheostomy: Is it a better option than bronchoscopic guided percutaneous tracheostomy? Med J Armed Forces India. 2015 Apr;71(2):158-64. doi: 10.1016/j.mjafi.2015.01.013. Epub 2015 Mar 12. PMID 25859079
- [Background] Gobatto AL, Besen BA, Tierno PF, Mendes PV, Cadamuro F, Joelsons D, Melro L, Park M, Malbouisson LM. Comparison between ultrasound- and bronchoscopy-guided percutaneous dilational tracheostomy in critically ill patients: a retrospective cohort study. J Crit Care. 2015 Feb;30(1):220.e13-7. doi: 10.1016/j.jcrc.2014.09.011. Epub 2014 Sep 22. PMID 25306240
- [Background] Flint AC, Midde R, Rao VA, Lasman TE, Ho PT. Bedside ultrasound screening for pretracheal vascular structures may minimize the risks of percutaneous dilatational tracheostomy. Neurocrit Care. 2009 Dec;11(3):372-6. doi: 10.1007/s12028-009-9259-z. Epub 2009 Aug 13. PMID 19680824